CLINICAL TRIAL: NCT00359931
Title: Neural Modeling and Brain Imaging of Tinnitus
Brief Title: Brain Imaging of Tinnitus
Status: Completed | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060218; 06-DC-0218
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-03-07

CONDITIONS: Hearing Disorder
Keywords: Neural Networks; Mathematical Modeling; Auditory Processing; Tinnitis; Hearing Loss
MeSH Terms: conditions — Hearing Disorders; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
This study will use magnetic resonance imaging (MRI) to compare brain function in three groups of people: hearing-impaired people with tinnitus; hearing-impaired people without tinnitus; and people with normal hearing and without tinnitus. Also known as "ringing in the ears," tinnitus is the false sensation of sounds.

Adults between 30 and 65 years of age who meet the following criteria may be eligible for this study:

* Mild to moderate hearing loss who have experienced tinnitus daily for at least 1 year
* Mild to moderate hearing loss who have never or rarely experienced tinnitus
* Normal hearing who have never or rarely experienced tinnitus

Candidates are screened with a medical history and questionnaires.

Participants have a detailed hearing test to measure hearing and the nature of tinnitus. In a second visit, subjects have a brief physical examination, followed by MRI scanning. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the subject lies on a table that can slide in and out of the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The subject may be asked to lie still for up to 8 minutes at a time. During the MRI, the subject performs computer-based tasks that involve listening to sounds. Another hearing test is done after the MRI.

DETAILED DESCRIPTION:
Subjective tinnitus, the false perception of sound in the absence of an acoustic stimulus, occurs frequently as a consequence of noise-induced deafness. The purpose of this study is to investigate the brain sites and mechanisms underlying tinnitus using a combined mathematical modeling and functional brain imaging experimental approach. Although studies have focused on the neural bases of tinnitus, it is not known why tinnitus arises only in certain cases of hearing loss, and the contribution of different brain regions in tinnitus perception is poorly understood. This in turn, prevents the development of better studies and new treatment methods for tinnitus. The primary hypothesis is that a network of brain regions, from auditory processing areas to emotional processing areas, contributes to, and modulates, tinnitus perception. The brain imaging study will be used to study differences in the network of brain regions involved in listening and discriminating sounds for tinnitus sufferers as compared to a control group of subjects with similar hearing loss but without tinnitus. This comparison should permit the identification of brain regions most active in tinnitus. An age matched control group without hearing loss and tinnitus will be included to determine those effects due to hearing loss alone. The mathematical computational modeling will use a previously developed large-scale neural network model of auditory processing in the cerebral cortex, which will be modified to induce tinnitus via different neural mechanisms. The modeling study should allow us to evaluate the contribution of different cortical regions and mechanisms to tinnitus perception; some changes in the model will be more successful than others in inducing tinnitus and in matching simulated brain imaging data with experimental brain imaging data. The modeling study will use the same stimuli and experimental paradigm as the functional brain imaging study. Comparing the experimental and modeling results will provide hypotheses about the most likely mechanism mediating tinnitus. Together, the modeling and experimental studies will advance our knowledge of the brain regions and mechanisms underlying tinnitus.

ELIGIBILITY:
* INCLUSION CRITERIA:

Plus Tinnitus Plus Hearing loss subjects.

* Adults, between the ages of 30 to 65 years.
* Are able to hear and perceive sounds used in the experiment in the range 250 Hz to 2 KHz and have high-frequency sensorineural hearing loss beginning no lower than 2 KHz.
* In good health and not currently taking certain medications regularly (e.g. antidepressants, antiseizure medications, antipsychotics, etc.).
* Experience tinnitus daily.
* Have had non-pulsatile tinnitus for at least 1 year.
* Have bilateral or bilateral with unilateral dominance tinnitus.

Minus Tinnitus Plus Hearing loss subjects.

* Adults, between the ages of 30 to 65 years.
* Are able to hear and perceive sounds used in the experiment in the range 250 Hz to 2 KHz and have high-frequency sensorineural hearing loss beginning no lower than 2 KHz.
* In good health and not currently taking certain medications regularly (e.g. antidepressants, antiseizure medications, antipsychotics, etc.).
* Have never or rarely (i.e. transient episodes experienced by virtually everyone) experienced tinnitus.

Minus Tinnitus Minus Hearing loss subjects or normal volunteers.

* Adults, between the ages of 30 to 65 years.
* Have normal hearing.
* In good health and not currently taking certain medications regularly (e.g. antidepressants, antiseizure medications, antipsychotics, etc.).

EXCLUSION CRITERIA:

* Subjects who have pacemakers, aneurysm clips, metallic prostheses or shrapnel fragments.
* Subjects incapable of giving informed consent.
* Subjects with a positive pregnancy test.
* Children below the age of 18 years.
* Subjects with hyperacusis or misophonia (hyper-sensitivity to loud noises).
* Subjects with mood disturbances such as depression or anxiety.
* Subjects with a history of temporomandibular joint problems or who present symptoms of pain and tenderness of the temporomandibular joint on examination.

Subjects may be excluded for the following reasons that may cause difficulty with interpretation of the imaging data:

* Subjects with mental or physical illnesses, other than tinnitus that may cause problems with participation in the study.
* Subjects with current uncontrolled hypertension, or significant past history of cardiovascular disease and diabetes melitus.
* Subjects with a history of head trauma with loss of consciousness, epilepsy, seizures, a history of chemotherapy (neurotoxic or ototoxic) and other medical conditions that may alter cerebral functioning.
* Subjects who are taking or have a history of taking recreational drugs or alcoholism.
* Subjects with unilateral or asymmetrical hearing loss who have not had (or cannot provide documentation of) comprehensive neuro-otologic workup will be excluded.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-07-28; Study Completion 2016-03-07

PRIMARY OUTCOMES:
The primary hypothesis is that a network of brain regions, from auditory processing areas to emotional processing areas, contributes to, and modulates, tinnitus perception. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Barry Horwitz, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mirz F, Gjedde A, Sodkilde-Jrgensen H, Pedersen CB. Functional brain imaging of tinnitus-like perception induced by aversive auditory stimuli. Neuroreport. 2000 Feb 28;11(3):633-7. doi: 10.1097/00001756-200002280-00039. PMID 10718327
- [Background] Giraud AL, Chery-Croze S, Fischer G, Fischer C, Vighetto A, Gregoire MC, Lavenne F, Collet L. A selective imaging of tinnitus. Neuroreport. 1999 Jan 18;10(1):1-5. doi: 10.1097/00001756-199901180-00001. PMID 10094123
- [Background] Mirz F, Gjedde A, Ishizu K, Pedersen CB. Cortical networks subserving the perception of tinnitus--a PET study. Acta Otolaryngol Suppl. 2000;543:241-3. doi: 10.1080/000164800454503. PMID 10909031